CLINICAL TRIAL: NCT03932604
Title: A Prospective, Multicenter, Randomized Controlled Trial Comparing Atrial Sensing ON-mode of VDD Implantable Cardioverter Defibrillator(ICD) to Atrial Sensing OFF-mode of VDD ICD in Detecting Atrial Fibrillation(Smart-Control Study)
Brief Title: Atrial Sensing Capability for Better Detection of Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: SMC-2019-01-149-03
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-06

CONDITIONS: Implantable Cardioverter Defibrillator; Atrial Fibrillation; Cardiac Event; Cardiac Arrhythmia
MeSH Terms: conditions — Atrial Fibrillation; Cardiovascular Diseases; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: Patients are randomly assigned as atrial sensing ON or Off mode
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atrial sensing OFF mode (No Intervention): VDD-ICD programmed as atrial sensing Off mode
- Atrial sensing ON mode (Active Comparator): VDD-ICD programmed as atrial sensing ON mode
  Interventions: Device: Atrial sensing On mode

INTERVENTIONS:
Device: Atrial sensing On mode — Single lead VDD-ICD programmed as atrial sensing On mode.
  Arms: Atrial sensing ON mode

SUMMARY:
This prospective multi-center randomized controlled study aims to compare atrial fibrillation detection and inappropriate therapy according to activation of atrial sensing capability in patients with implantable cardioverter defibrillator.

DETAILED DESCRIPTION:
Implantable cardioverter defibrillators(ICD) therapy has been shown to reduce sudden cardiac death and improve survival in cardiac arrest survivors as well as in heart failure patients with left ventricular dysfunction.

Atrial fibrillation (AF) is commonly found in ICD implantation patients up to 50%. AF is an independent predictor of mortality, inappropriate shock, and embolic events. Therefore, early detection of AF in patients with ICD is essential for improving the quality of life and overall prognosis of the patients.

Conventional ICDs consist of a single chamber (SC) ICD with a lead only in the right ventricle (RV) and dual chamber (DC) ICD with each lead in the right atrium (RA) and RV. SC ICD has the advantage of shorter procedure time, lower cost compared to DC ICD. In contrast, DC ICD has the advantage of being able to monitor atrial arrhythmic events, but complication rates were higher and additional cost and longer procedure time are usually required than SC ICD. Sixty percent of ICD implantation patients who have are SC ICD Recently, a unique ICD lead with atrial sensing ring capable of monitoring the atrial electrical signals has been developed [Intica 7 VR-T DX ICD (Biotronik., Germany)]. Therefore, turning off the atrial sensing function makes it functionally the same as SC ICD whereas turning on makes it function similar to DC ICD without additional cost and procedure time.

Therefore, Detection of AF could be made earlier with VDD ICD versus conventional SC ICD without atrial sensing capability, providing a better chance to improve the prognosis of ICD patients. However, no study exists which shows whether VDD ICD is better for detecting atrial tachyarrhythmia than conventional SC ICD. Therefore, we designed a multicenter prospective randomized study comparing the AF diagnostic efficacy of VDD ICD (with atrial sensing 'ON') against conventional SC ICD. As the second phase, we also plan to compare inappropriate therapy rate according to atrial sensing status of VDD ICD.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 19 years
2. indication for ICD implantation according to guidelines
3. atrial fibrillation didn't detect by electrocardiogram or Holter test within the past 1 year from the ICD implantation, and
4. CHA2DS2VASc score ≥1 point in male or ≥ 2 in female

Exclusion Criteria:

1. persistent or permanent atrial fibrillation (AF)
2. atrial fibrillation detected by electrocardiogram or Holter test within the past 1 year from the ICD implantation
3. history of the catheter or surgical ablation of AF or taking antiarrhythmic drug
4. scheduled to undergo heart transplant within 1 year
5. life expectancy < 1 year
6. requiring atrial pacing

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | from enrollment to last follow-up (2 years)
  cardiac implantable electronic device-detected or clinical atrial fibrillation
Inappropriate device therapy | from enrollment to last follow-up (2 years)
  inappropriate ATP or shock

SECONDARY OUTCOMES:
Number of Participants with complications associated with atrial fibrillation | from enrollment to last follow-up (2 years)
  thromboembolic events, heart failure
Number of Participants with ventricular arrhythmia | from enrollment to last follow-up (2 years)
  cardiac implantable electronic device-detected or clinical ventricular arrhythmia
Number of Participants with major adverse composite events | from enrollment to last follow-up (2 years)
  cardiac death, all cuase death, stroke, atrial fibrillation or flutter, ventricular tachyarrhythmia, hospitalization for heart failure
atrial lead sensing stability | from enrollment to last follow-up (2 years)
  Atrioventricular synchrony ratio

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, PhD, Principal Investigator — Samsung Medical Center
Locations (28):
- South Korea (28):
  - Sejong General Hospital, Bucheon-si
  - Inje University Busan Paik Hospital, Busan
  - Samsung Changwon Medical Center, Changwon
  - Chungbuk National University Hospital, Cheongju-si
  - Kangwon National University Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeongnam University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - GangNeung Asan Hospital, Gangneung
  - National Health Insurance Service Ilsan Hospital, Goyang
  - Gachon University, Donginchoen Gil Hospital, Incheon
  - Inha University Hospital, Incheon
  - Mediplex Sejong Hospital, Incheon
  - Kosin University Gospel Hospital, Pusan
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Hallym University Medical Center-Kangnam, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - Koera University Guro Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - VHS Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gwag HB, Kim HR, Park SJ, Kim J, Chung TW, Choi JH, Kim JY, Park KM, On YK, Kim JS. The efficacy of single-lead implantable cardioverter-defibrillator with atrial sensing dipole to detect atrial fibrillation and to reduce inappropriate therapy according to atrial sensing ON or OFF: Rationale and design of the SMART-CONTROL study, a prospective multicenter randomized trial. Am Heart J. 2022 Sep;251:25-31. doi: 10.1016/j.ahj.2022.05.008. Epub 2022 May 12. PMID 35568193